CLINICAL TRIAL: NCT03950245
Title: Importance of Endogenous Glucagon-like Peptide-1 and Glucose-dependent Insulinotropic Polypeptide for Postprandial Glucose Metabolism After Roux-en-Y Gastric Bypass and Sleeve Gastrectomy Surgery
Brief Title: Incretin Hormone Antagonism After Bariatric Surgery
Acronym: INCA-BAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Morten Gadegaard Hindsø, MD, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MH-INKA-BAR-19
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Bariatric Surgery
Keywords: glucagon-like peptide-1; glucose-dependent insulinotropic polypeptide; Roux-en-Y gastric bypass; sleeve gastrectomy; gastric bypass; bariatric surgery; glucose; diabetes; exendin(9-39); GIP(3-30)
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastric bypass operated patients (Other): Four test days in a randomized, patient-blinded, cross-over design
  Interventions: Other: Placebo; Other: GLP-1 antagonism; Other: GIP antagonism; Other: GLP-1 and GIP antagonism
- Sleeve gastrectomy operated patients (Other): Four test days in a randomized, patient-blinded cross-over, design
  Interventions: Other: Placebo; Other: GLP-1 antagonism; Other: GIP antagonism; Other: GLP-1 and GIP antagonism
- Un-operated controls (Other): Four test days in a randomized, patient-blinded cross-over, design
  Interventions: Other: Placebo; Other: GLP-1 antagonism; Other: GIP antagonism; Other: GLP-1 and GIP antagonism

INTERVENTIONS:
Other: Placebo — Four-hour liquid mixed meal tests and a subsequent ad libitum meal during saline infusion.
Other: GLP-1 antagonism — Four-hour liquid mixed meal tests and a subsequent ad libitum meal during exendin 9-39 and saline infusion.
Other: GIP antagonism — Four-hour liquid mixed meal tests and a subsequent ad libitum meal during GIP(3-30) and saline infusion.
Other: GLP-1 and GIP antagonism — Four-hour liquid mixed meal tests and a subsequent ad libitum meal during exendin and GIP(3-30) infusion.

SUMMARY:
Using the glucagon-like peptide-1 (GLP-1) antagonist exendin(9-39) and the glucose-dependent insulinotropic peptide (GIP) antagonist GIP(3-30), the purpose of this study is to clarify the importance of endogenous GLP-1 and GIP for postprandial glucose metabolism after RYGB and SG in subjects with normal glucose tolerance. We hypothesize that GLP-1 is more important after RYGB, and GIP is more important after SG, for postprandial glucose tolerance and beta-cell function. A group of un-operated subjects with normal glucose tolerance will serve as controls.

ELIGIBILITY:
Inclusion Criteria, surgery groups:

* Age > 18 years
* RYGB or SG operation > 12 months prior to inclusion
* Weight stable (± 3 kg during the last month)
* HbA1c < 48 mmol/mol before surgery, and no history of diabetes
* HbA1c < 48 mmol/mol and fasting plasma glucose < 6.1 mmol/l at inclusion

Inclusion Criteria, control group:

* Age > 18 years
* no former RYGB- or SG operation
* Weight stable (± 3 kg during the last month)
* HbA1c < 48 mmol/mol, fasting plasma glucose < 6.1 mmol/l and no history of diabetes

Exclusion Criteria:

* Thyrotoxicosis or inadequately treated hypothyreosis
* Hemoglobin < 6.5 mmol/l at inclusion
* Pregnancy or breast feeding
* Medication affecting the planned examinations

Matching between groups

* Age
* Sex
* BMI at inclusion and for surgery groups also pre-surgery BMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
iAUC glucose | 240 minutes
  Main comparison between groups: delta iAUC glucose (iAUC exendin(9-39) test day - iAUC GIP(3-30) test day) in the RYGB group compared to the SG group

SECONDARY OUTCOMES:
Beta-cell glucose sensitivity (β-GS) | 240 minutes
  Main comparison between groups: delta β-GS (β-GS exendin(9-39) test day - β-GS GIP(3-30) test day) in the RYGB group compared to the SG group

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine N Bojsen-Møller, MD, PHD, Principal Investigator — Dept. of Endocrinology, Hvidovre Hospital, Denmark; Morten G Hindsø, MD, Principal Investigator — Dept. of Endocrinology, Hvidovre Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department of Endocrinology, Hvidovre
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No